CLINICAL TRIAL: NCT00529893
Title: Efficacy of Atomoxetine in the Neuropsychological Tests Among Children With ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 200612093M
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2013-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention-deficit/Hyperactivity Disorder; neuropsychological functioning; Atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is examine the efficacy of atomoxetine on executive functioning measures including the Continuous Performance Test (CPT) and the executive function measures of the Cambridge Automated Neuropsychological Test Automated Battery (CANTAB).

DETAILED DESCRIPTION:
The rationale of this proposal is based upon the high prevalence (7.5% in Taiwan (Gau et al., 2004b)), the magnitude of the short- and long-term impact on individuals, family, and society, the responsibility of attention-deficit hyperactivity disorder ADHD to treatments with CNS stimulants and Atomoxetine. Although numerous studies have shown that methylphenidate demonstrates significant effect on improving neuropsychological functioning including inhibition of executive function (e.g., Aron et al., 2003; Kempton et al., 1999; Konrad et al., 2004) and motor control measures (e.g., Moll et al., 2000), there has been no study examining the effect of Atomoxetine on the improvement of response inhibition or other neuropsychological functioning among children with ADHD. As several clinical trials have shown the efficacy of Atomoxetine in improving the core symptoms of ADHD (e.g., Eiland and Guest, 2004; Michelson et al., 2002) and Atomoxetine has been approved by FDA as first line medication for child and adult ADHD in 2002, we anticipate that Atomoxetine will demonstrate significant efficacy on treating ADHD by improvement of neuropsychological measures.

The objectives of this study are:

1. To examine the efficacy of atomoxetine on executive functioning measures including the Continuous Performance Test (CPT) and the executive function measures of the Cambridge Automated Neuropsychological Test Automated Battery (CANTAB).
2. To examine the efficacy of atomoxetine on other neuropsychological measures including the Wisconsin Card Sorting Test (WCST), and the attention, memory, and paired learning tests of the CANTAB.
3. To validate the ADHD using psychopathological, neuropsychological, functional brain imaging, behavioral, and social correlates.

This study is an open label, non randomized, clinical trial with daily dose of atomoxetine 1.2 mg/kg for subjects with ADHD. Thirty drug-naïve children with DSM-IV ADHD and 30 normal children matched in sex, age, and IQ will be recruited. All of the participants will be assessed by the CPT, WSCT, CANTAB, and several measures covering domains of ADHD symptoms and social functioning. Subjects with ADHD will be reassessed using the neuropsychological tests and other measures on Week 4 (Visit 2) 3 days, Week 12 (Visit 2) 3 days of treatment with atomoxetine 1.2 mg/kg.

The sample will consist of 30 subjects with ADHD, aged 10 to 15, and 30 subjects without ADHD, who are matched in age, sex, and IQ as cases. We anticipate that this study will provide enough evidence to support the efficacy of Atomoxetine not only on the symptoms improvement but also neuropsychological measures and fMRI studies among children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

(1) subjects had the clinical diagnosis and the K-SADS-E of DSM-IV ADHD; (2) their ages range from 10 to 15; (3) subjects must not have taken any medication used to treat ADHD; (4) subjects' IQ should be larger than 80; (5) subjects and their parents and teachers consent to participate and have the ability to complete self-administered measures in this study.

Exclusion Criteria:

The subjects will be excluded from the study if they currently meet criteria or have a history of the following conditions as defined by DSM-IV: Shizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, Pervasive Developmental Disorder, Anxiety Disorders, Phobia, Obsessive-Compulsive Disorder, Depressive Disorders, or Bipolar Disorders. In addition, subjects will be excluded from this study if any evidence showing medical problems, or seizure. Moreover, the subjects will be excluded from the control group if have a history of the following condition as defined by DSM-IV: ADHD, ODD, or CD in addition to the above exclusion criteria.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects are diagnosed as DSM-IV, Attention Deficit Hyperactivity Disorder (ADHD).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The Efficacy of Once-Daily Atomoxetine Hydrochloride on Executive Function in Taiwanese Children with Attention-deficit/ Hyperactivity Disorder | 12 weeks
  Patients with ADHD performed worse in the backward digit span task, CPT, IED and RVIP than the controls. Their significant improvement in executive function after treatment with atomoxetine for 4 weeks included fewer omission and commission errors, fewer hit reaction time standard errors, and less variability in the CPT; fewer total errors and trials in the IED; higher probability of hits, total correction rejection, and total hits, fewer total misses, and shorter latency in the RVIP; longer span length and fewer total usage errors in the SSP; fewer errors and strategy utilization in the SWM; and more problems solved, fewer mean moves, and shorter subsequent thinking time in the SOC. Atomoxetine significantly reduced ADHD-related symptoms over time.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Gau SS, Shang CY. Improvement of executive functions in boys with attention deficit hyperactivity disorder: an open-label follow-up study with once-daily atomoxetine. Int J Neuropsychopharmacol. 2010 Mar;13(2):243-56. doi: 10.1017/S1461145709990836. Epub 2009 Oct 23. PMID 19849892